CLINICAL TRIAL: NCT06989853
Title: Advancing Troiluzole as a Treatment for Methamphetamine Use Disorder: A Human Laboratory Study
Brief Title: Methamphetamine and Troriluzole
Acronym: BED IN 46
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 99084; R01DA060632 (NIH)
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Use Disorder
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will be treated daily with an oral placebo.
  Interventions: Drug: Placebo
- Troriluzole Dose 1 (Experimental): Subjects will be treated daily with oral troriluzole (140 mg).
  Interventions: Drug: Placebo; Drug: Methamphetamine
- Troriluzole Dose 2 (Experimental): Subjects will be treated daily with oral troriluzole (280 mg).
  Interventions: Drug: Placebo; Drug: Methamphetamine

INTERVENTIONS:
Drug: Placebo — The effects of placebo will be determined.
Drug: Methamphetamine — Placebo and methamphetamine will be administered intravenously during experimental sessions.
  Arms: Troriluzole Dose 1; Troriluzole Dose 2

SUMMARY:
This will be a human laboratory study evaluating the influence of troriluzole treatment on the effects of methamphetamine. Supported by and included in the Helping to End Addiction Long-term® (HEAL) Initiative.

ELIGIBILITY:
Inclusion Criteria:

1. able to speak/read English,
2. not seeking treatment for drug use at the time of the study,
3. female or male between the ages of 18 and 55 years,
4. recent methamphetamine use verified by methamphetamine positive urine, as well as fulfillment of DSM-5 diagnostic criteria for MUD,
5. judged to be medically and psychiatrically healthy by study physicians other than the diagnosis for MUD (and OUD for the co-morbid MUD and OUD group, see below) at the time of screening,
6. ECG, read by a cardiologist, within normal limits,
7. females using an effective form of birth control and not pregnant or breastfeeding,
8. no known contraindications (e.g., hepatic disease [save for asymptomatic HCV status as cleared by study physician]) or allergies to troriluzole. Individuals in the MUD and OUD group must also report recent opioid use, verified by opioid positive urine, as well as fulfillment of DSM-5 diagnostic criteria for OUD with physiologic dependence (determined to not be physically dependent if a participant arrives with a urine sample for drug screening that is negative for a short-acting opioid and does not have a score of 5 or greater on the clinical opioid withdrawal scale [COWS]).

Exclusion Criteria:

1. unable to speak/read English,
2. seeking treatment for drug use,
3. under 18 years or over 55 years,
4. no recent methamphetamine use as indicated by methamphetamine negative urine and no DSM-5 diagnosis of MUD,
5. judged to be medically and psychiatrically unhealthy by study physicians at the time of screening,
6. ECG, read by a cardiologist, outside normal limits,
7. females not using an effective form of birth control or pregnant or breastfeeding,
8. blood pressure readings indicative of hypertension (i.e., blood pressure > 140/90 mmHg) on 2 consecutive screening visits,
9. BMI < 18 or > 30; weight < 50 kg,
10. taking any medications prescribed by a physician for a chronic condition,
11. any laboratory chemistry values (e.g., LFTs) > 3 times normal at screening or during admission,
12. history of serious physical disease or diagnosis of any disorder (e.g., current hepatic disease [save for asymptomatic HCV status; as noted above], histories of seizure, diabetes, asthma or CNS tumors) or current or past histories of psychiatric disorder, including current or recent suicidal ideation that would limit compliance in the study, other than MUD or tobacco use disorder (and OUD for the co-morbid MUD/OUD group only) that in the opinion of the study physicians would interfere with participation and
13. contraindications (e.g., hepatic disease) or allergies to troriluzole.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Reinforcing Effects of Methamphetamine | 9 times over approximately 1 month inpatient admission
  Number of Times Subjects Hypothetically Choose Methamphetamine Over Money between $0 and $140

CONTACTS AND LOCATIONS:
Locations (1):
- Psychopharmacology of Addiction Laboratory, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
All data from this project will be preserved and shared through an NIH-funded repository. Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 02/28/2029 (anticipated); available in perpetuity
Access Criteria: investigators working under an institution with a Federal Wide Assurance (FWA)